CLINICAL TRIAL: NCT04321005
Title: Surgical Safety and Effectiveness in Orthopedics: Swiss-wide Multicenter Evaluation and Prediction of Core Outcomes in Arthroscopic Rotator Cuff Reconstruction
Acronym: ARCR_Pred
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other); Swiss Orthopaedics (Unknown); Schweizerische Versicherungsanstalt (SUVA) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019-02076; ch20Mueller
Record Dates: First submitted 2020-03-03; First posted 2020-03-25 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Rotator Cuff Tear
Keywords: Oxford Shoulder Score (OSS); shoulder stiffness; arthroscopic rotator cuff repair
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: arthroscopic rotator cuff reconstruction — arthroscopic rotator cuff reconstruction and assessment with evaluation and prediction of core outcomes

SUMMARY:
Surgical safety and effectiveness in orthopedics: Swiss-wide multicenter evaluation and prediction of core outcomes in arthroscopic rotator cuff reconstruction.

DETAILED DESCRIPTION:
In this project prospective data are collected from a representative group of specialized clinics performing arthroscopic rotator cuff repair (ARCR) to serve as reference baseline and outcome values, as well as the development of prediction models for individual patients.

Ultrasound and MRI (on a subset of patients) examination will be performed at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* diagnosed with a partial or full-thickness rotator cuff tear using magnetic resonance imaging (MRI)
* planned primarily surgical partial or complete repair by arthroscopic procedure
* able to understand the content of the patient information/ consent form and give consent to take part in the project

Exclusion Criteria:

* surgical procedure for irreparable tears, i.e. muscle transfer, acromio-humeral spacer or superior capsular reconstruction
* revision surgery (prior repair of the rotator cuff in the same shoulder)
* planned open or mini-open reconstructions
* patients with a language barrier hindering questionnaire completion (either in German, French, Italian or English)
* patients unlikely to attend clinical follow-up
* pregnancy
* legal incompetence

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated for a partial or full-thickness rotator cuff tear with primarily surgical partial or complete repair by arthroscopic procedure
Sampling Method: Probability Sample
Enrollment: 973 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Patient-reported change in shoulder functional outcome OSS | at Baseline and at 6 months after surgery.
  The Oxford Shoulder Score (OSS) is a condition-specific questionnaire developed for patients with a degenerative or inflammatory state of the shoulder. It contains twelve items to be answered by the patient independently, which deal with pain (degree, time point) and possible handicaps in private and professional life.
  There are five categories of response for every question, corresponding to a score ranging from 0 to 4. Scores are combined to give a single score, with a range from 0 (worst outcome) to 48 (best outcome).
Change of shoulder stiffness | at Baseline and at 6 months after surgery.
  this event was defined as a postoperative restriction in passive shoulder motion diagnosed within 6 months after ARCR in at least two of the motion planes of flexion, abduction and external rotation in 0° abduction. Motion restriction is to be assessed separately for each plane

SECONDARY OUTCOMES:
Local AEs (Adverse events) according to the ARCR Core Event Set (CES) | 24 months
  * Recurrent defect of repaired tendon(s) at 12 months: at least one repaired tendon is diagnosed with a recurrent defect by ultrasound examination.- Persistent or worsening pain
  * Infection
  * Any local event
Constant Murley Score (CMS) | at 6 and 12 months
  The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient. The scale is from 1 to 100 with higher scores indicating better outcome.
Shoulder strength (kg) in abduction at 6 and 12 months | at 6 and 12 months
  Highest possible Weight load of the Shoulder measured by dynamometer
Change in Patient-reported shoulder pain on a Numeric Rating Scale (NRS) | at 6, 12 months and 24 months
  The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults.
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. A Higher Score means a worse outcome. The common format is a horizontal bar or line. Similar to the VAS, the NPRS is anchored by terms describing pain severity extremes.
Change in Oxford Shoulder Score (OSS) | at 6, 12 months and 24 months
  The Oxford Shoulder Score (OSS) is a validated patient-reported outcome measure (PROM). It's a shoulder-specific instrument designed to assess the outcome of all shoulder surgeries (with the exception of instability surgery). The combined total gives a minimum score of 12 and a maximum of 60. Higher scores in the OSS imply worse functionality while lower scores imply better functionality.
Subjective Shoulder Value (SSV) | at 6, 12 months and 24 months
  The SSV is defined as a patient's subjective shoulder assessment expressed as a percentage of an entirely normal shoulder, which would score 100%
Nonrestorative sleep (NRS) to assess Patient-reported quality of sleep | at 6, 12 and 24 months
  Nonrestorative sleep (NRS) is defined as the subjective experience that sleep has not been sufficiently refreshing or restorative. On a scale from 0-10, 0 is best possible outcome measure and 10 is worst possible outcome measure.
Return to work, change of working condition | at 6, 12 and 24 months
  Return to work, change of working condition is measure in a standardized questionnaire noting among others absences
PROMIS Depression and Anxiety Short Formto assess level of depression and anxiety | at 6, 12 and 24 months
  Measured by Patient-Reported Outcomes Measurement Information System (PROMIS) scores. For PROMIS measures, higher scores equals more of the concept being measured.
Patient perceived shoulder functionality change, acceptability of own symptom state | at 6, 12 and 24 months
  Patient perceived shoulder functionality change, acceptability of own symptom state are measured with emphasis on minimally clinically important differences as stated in the cited literature with the according scored measurements
Quality of life (utilities and general health): EQ-5D-5L | at 12 and 24 months
  Measured through EuroQoL version (EQ-5D-5L). The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. This tool has an overall health scale where the rater selects a number between 1-100 to describe the condition of their health, 1 being the worst and 100 being the best possible outcome.
Adverse event (AE) assessment: AEs reported by clinicians and patients | 6 months
  AEs reported by clinicians and patients (including non-local AEs within 6 months after surgery) b. Final independent surgeon and patient-rated assessment of AEs according to perceived severity and relation to treatment (according to perceived severity (rating scale from 0 [no complication] to 100 [death] [67]) and disturbance) c. Comprehensive Complication Index (CCI)
Adverse event (AE) assessment: Final independent surgeon and patient-rated assessment of AEs | 6 months
  Final independent surgeon and patient-rated assessment of AEs according to perceived severity and relation to treatment (according to perceived severity (rating scale from 0 [no complication] to 100 [death]) and disturbance)
Adverse event (AE) assessment:Comprehensive Complication Index (CCI) | 6 months
  Comprehensive Complication Index (CCI): The Comprehensive Complication Index is based on the complication grading by Clavien-Dindo Classification and implements every occurred complication after an intervention. The overall morbidity is reflected on a scale from 0 (no complication) to 100 (death).
Rotator cuff and biceps tendon integrity by MRI | at 12 months
  Postoperative integrity status of the rotator cuff classified by MRI
Rotator cuff muscle fatty infiltration by MRI | at 12 months
  Rotator cuff muscle fatty infiltration by MRI
Status of repair implants e.g. anchors by MRI | at 12 months
  Status of repair implants e.g. anchors by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Müller, PD Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (20):
- Department for Shoulder and Elbow surgery Center for Musculoskeletal Surgery Campus Virchow, Berlin, Germany
- Switzerland (19):
  - Kantonsspital Baden AG,, Baden, Aarau
  - Kantonsspital Baselland, Binningen, Basel-Landschaft
  - Hirslanden Klinik Birshof, Münchenstein, Basel-Landschaft
  - Klinik tür Orthopädische Chirurgie und Traumatologie des Bewegungsapparates Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Zentrum für Orthopädie & Neurochirurgie In-Motion, Wallisellen, Canton of Zurich
  - Klinik Gut, St. Moritz, Kanton Graubünden
  - Hopital du Valois (RSV), Martigny-Ville, Valais
  - University Hospital Basel, Basel
  - ARTHRO Medics AG, Basel
  - Sonnenhof, Bern
  - Inselspital, Bern
  - Hirslanden Clinique de Colline, Geneva
  - University Hospital Geneva, Geneva
  - Regional Hospital Lugano, Lugano
  - Bürgerspital Solothurn, Klinik für Orthopädie und Traumatologie, Solothurn
  - Kantonsspital Winterthur, Klinik für Orthopädie und Traumatologie, Winterthur
  - Schulthess Klinik, Zurich
  - Universitätsklinik Balgrist, Zurich
  - Endoclinic, Zurich

REFERENCES:
- [Derived] Audige L, Bucher HCC, Aghlmandi S, Stojanov T, Schwappach D, Hunziker S, Candrian C, Cunningham G, Durchholz H, Eid K, Flury M, Jost B, Ladermann A, Moor BK, Moroder P, Rosso C, Schar M, Scheibel M, Spormann C, Suter T, Wieser K, Zumstein M; ARCR_Pred Study Group; Muller AM. Swiss-wide multicentre evaluation and prediction of core outcomes in arthroscopic rotator cuff repair: protocol for the ARCR_Pred cohort study. BMJ Open. 2021 Apr 22;11(4):e045702. doi: 10.1136/bmjopen-2020-045702. PMID 33888530